CLINICAL TRIAL: NCT06640283
Title: Dynamic Assessment of ctDNA in Patients With Cervical and Anal Canal Tumors to Optimize Follow-up and Clinical Outcomes in the Brazilian Unified Health System (SUS)
Brief Title: Dynamic ctDNA Assessment in Cervical and Anal Canal Tumors: Optimizing Follow-up and Clinical Outcomes
Acronym: ANA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Maria del Pilar Estevez Diz, Oncologist, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP5125/2024; 79795024.8.0000.0068 (Registry Identifier: Certificate of Ethical Review Submission); 444027/2023-8 (Other Grant/Funding Number: CNPq)
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: HPV-Related Carcinoma; Uterine Cervical Cancer; Anal Canal Cancer; HPV-Related Anal Squamous Cell Carcinoma; HPV-Related Cervical Carcinoma
Keywords: HPV; ctDNA; Cervical tumors; Anal canal tumors; Molecular diagnosis; Diagnostic test; Biomarkers
MeSH Terms: conditions — Uterine Cervical Neoplasms; Anal Canal Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: 84 to150 patients will be tested for HPV in their tumor samples 68 patients with negative ctDNA after CRT will be monitored with ctDNA plus routine image 16 patients with positive ctDNA after CRT will receive anti-PD1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active laboratory monitoring (Other): Phase I Monitoring through collection of laboratory tests
  Interventions: Diagnostic Test: ctDNA test
- Intervention with Immunotherapy (Experimental): Phase II for participants who are ctDNA positive after standard treatment.
  Intervention will be with Pembrolizumab
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Diagnostic Test: ctDNA test — ctDNA involves the collection of peripheral blood samples for the analysis of circulating tumor DNA (ctDNA). The samples are processed using next-generation sequencing (NGS) and/or digital polymerase chain reaction (PCR) techniques to detect specific genetic alterations related to the tumor. The objective is to assess the presence and quantity of ctDNA, providing information on tumor burden and treatment response.
  Arms: Active laboratory monitoring
Drug: Pembrolizumab — Participants will receive the institution's standard treatment during Phase I. If ctDNA remains positive between 8 and 12 weeks after the standard treatment, the participant will be invited to proceed to Phase II, which will consist of intravenous immunotherapy for up to 12 months, or until disease progression or unacceptable toxicity occurs. Continuous monitoring with ctDNA testing will be performed during Phase II.
  Arms: Intervention with Immunotherapy

SUMMARY:
After definitive radiotherapy (RT) treatment (with or without chemotherapy), cervical and anal canal neoplasms frequently exhibit disease persistence or recurrence. Due to the local inflammatory process post-treatment, response assessment by imaging (current gold standard) is limited, often necessitating multiple follow-ups and repeated invasive biopsies. Conventional follow-up is complex and costly, requiring equipment from secondary and tertiary services, trained radiologists, and patient exposure to radiation and contrast.

In this context of human papillomavirus(HPV)-related neoplasms, recent studies have demonstrated the role of ctDNA (circulating tumor DNA) in assessing the risk of recurrence or disease progression, providing a rationale for using the tool in two fronts:

* Optimizing follow-up based on serial monitoring of ctDNA;
* Selecting patients with positive ctDNA after RT, who are at high risk of recurrence, for treatment intensification.

Monitoring with ctDNA as a standalone follow-up tool in cases evolving with negative ctDNA after RT has the potential to replace imaging exams, being a minimally invasive test performed on a peripheral blood sample. Currently, ctDNA testing has expensive methodologies not available in the Unified Health System (SUS). This project aims to develop a methodology for ctDNA evaluation focused on HPV ctDNA research that is low-cost and executable in SUS, as well to assess the accuracy of this test in the population with HPV-related tumors.

Additionally, we will evaluate whether the early introduction of immunotherapy in patients with positive ctDNA after definitive treatment can increase cure rates. Immunotherapy already has a well-defined role in the treatment of metastatic HPV-related neoplasms. Recently, the use of anti-programmed death-1 (anti-PD1) has also shown benefits in patients with locally advanced cervical cancer with a high risk of recurrence who are candidates for chemoradiotherapy (CRT). Therefore, its use focused on HPV-related tumors, as well as a better understanding of which patients benefit from this strategy, warrants further investigation.

DETAILED DESCRIPTION:
The ANA study is a research project aimed at enhancing the treatment and outcomes for patients with cervical and anal canal cancer by using innovative diagnostic and therapeutic methods. The study consists of the following phases:

* Patient identification and selection;
* Recruitment of patients diagnosed with cervical or anal canal cancer who are candidates for treatment with radiotherapy (RT), with or without chemotherapy: patients will be selected based on specific criteria to ensure a representative cohort;
* Development and validation of the ctDNA HPV Test: development of a sensitive and specific test to detect HPV DNA in the blood. This test will undergo rigorous validation to ensure its accuracy and reliability;
* ctDNA monitoring: blood samples collection from patients during treatment and follow-up. ctDNA levels will be monitored in real-time to early detection of residual or recurrent disease. This non-invasive method aims to provide a more accurate assessment of treatment efficacy and disease progression. The results of ctDNA will be compared with traditional imaging methods.
* Complementary immunotherapy treatment: patients with positive ctDNA results after (chemo)radiotherapy will be considered for additional immunotherapy. This phase will evaluate the benefits of combining immunotherapy with standard (chemo)radiotherapy in order to improve patient outcomes;
* Follow-up and outcome evaluation: long-term follow-up of patients to assess clinical outcomes, including survival and quality of life.

The ANA study aims to set new standards in the follow-up and management of HPV-related cervical and anal canal cancer by improving patient care within the Brazilian public health system (SUS).

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of anal canal or cervical cancer.
2. Documented presence of HPV.
3. Locally confined or locally advanced disease, defined as:

   1. Anal canal carcinoma stage I to III, according to American Joint Committee on Cancer (AJCC) 8th edition;
   2. Cervical carcinoma stage I B2 to IV A, according to AJCC 8th edition.
4. Indication for definitive treatment with radiotherapy, with or without concomitant chemotherapy.
5. Eastern Cooperative Oncology Group (ECOG)-Performance Status (PS) 0 - 1.
6. Age ≥ 18 years.
7. Signing of the Informed Consent Form (ICF).
8. HIV-positive patients may be included if Cluster of Differentiation 4(CD4) count is greater than or equal to 200.
9. Patients may participate in other concurrent studies, as long as they do not involve interventions related to the treatment of the underlying cancer.

Exclusion Criteria:

1. Patients with unequivocal distant metastasis at diagnosis.
2. For participants with positive ctDNA after treatment, those candidates for participation in Phase II will be excluded if there is unequivocal radiological progression in the first imaging exam after the completion of radiotherapy (with or without chemotherapy) or routine indication for salvage surgery immediately after the conclusion of definitive treatment.
3. Need for recurrent blood transfusions, such as weekly frequency.
4. Another uncontrolled disease representing a life risk, as determined by medical judgment.
5. Personal history of another active invasive malignant neoplasm in the last 5 years, except for non-melanoma skin carcinomas and in situ carcinomas.
6. Pregnant individuals.
7. Active opportunistic infection or disease.
8. History of autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
General Objective | 2 years
  The objective of this study is to develop and validate a low-cost ctDNA test focused on detecting HPV-associated ctDNA for use in patients within the Brazilian Unified Health System (SUS). The test will be evaluated for its effectiveness in improving traditional monitoring methods and guiding the intensification of adjuvant treatment for anogenital neoplasms, including anal canal and cervical cancer. The impact of the test will be measured by correlating ctDNA detection with clinical outcomes of patients over time.

OTHER OUTCOMES:
Number of HPV-focused ctDNA tests developed and validated | 2 years
  Measure the number of HPV-related ctDNA tests developed and validated for detecting HPV ctDNA in patients with anogenital neoplasms.
Performance of the validated HPV-related ctDNA test | 2 years
  Measure the accuracy and specificity of the validated HPV-related ctDNA test, including the assessment of HPV typing, ctDNA, and HPV E6*I messenger ribonucleic acid (mRNA) levels in the study population.
Comparison of accuracy between standard ctDNA and HPV-focused ctDNA | 2 years
  valuate the accuracy of standard ctDNA compared to HPV-focused ctDNA and in relation to standard radiological control, based on routine imaging, through serial testing of ctDNA and HPV ctDNA after completion of treatment with definitive radiotherapy or chemoradiotherapy.
Comparison with Commercially Available HPV ctDNA Tests | 2 years
  Compare the diagnostic accuracy of standard ctDNA with HPV-focused ctDNA and standard radiological control, using routine imaging and serial ctDNA tests after definitive treatment with radiotherapy or chemoradiotherapy.
Comparison of performance between the locally developed HPV ctDNA test and commercially available tests | 2 years
  Compare the sensitivity, specificity, and overall performance of the locally developed HPV ctDNA test with commercially available tests on the market.
Direct costs of the ctDNA test | 2 years
  Measurement of the costs associated with performing the ctDNA test, including materials, labor, and technology used.
Disease progression reduction rate with the use of immunotherapy | 2 years
  Measure the rate of disease progression reduction in patients with positive ctDNA after definitive treatment, in response to the use of immunotherapy.
Influence of PD-L1 expression and HPV type on immunotherapy response | 2 years
  Relationship between PD-L1 expression levels and HPV types on the immunotherapy response in patients with positive ctDNA. PD-L1 levels will be quantified using immunohistochemistry, and the HPV types present in tumor samples will be categorized. The outcomes will include the treatment response rate and progression-free survival, recorded over a two-year period.
Correlation between PD-L1 expression and HPV type with immunotherapy response | 2 years
  Measure the correlation between PD-L1 expression and HPV type with the response rate to immunotherapy in patients with positive ctDNA, quantifying the impact of these variables on the effectiveness of immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Maria DP Estevez Diz, Doctor, Principal Investigator — Oncologist
Locations (1):
- Instituto do Câncer do Estado de São Paulo - ICESP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
It has been decided not to share individual participant data (IPD) related to the study for several reasons. Protecting the privacy of participants is a priority. Sharing IPD may expose sensitive information that, even when de-identified, can be traced back to individuals.
  Furthermore, the complexity of the data makes sharing challenging without the risk of misunderstandings or misinterpretations, which could compromise the integrity of the research. Sharing IPD without the explicit consent of participants may violate ethical principles of respect and protection.
  There is also a need to comply with regulatory guidelines governing data sharing to avoid potential legal issues. Finally, the focus will be on disseminating aggregated results that can benefit the scientific community and the public without compromising individual privacy.

REFERENCES:
- [Background] Bernard-Tessier A, Jeannot E, Guenat D, Debernardi A, Michel M, Proudhon C, Vincent-Salomon A, Bieche I, Pierga JY, Buecher B, Meurisse A, Francois E, Cohen R, Jary M, Vendrely V, Samalin E, El Hajbi F, Baba-Hamed N, Borg C, Bidard FC, Kim S. Clinical Validity of HPV Circulating Tumor DNA in Advanced Anal Carcinoma: An Ancillary Study to the Epitopes-HPV02 Trial. Clin Cancer Res. 2019 Apr 1;25(7):2109-2115. doi: 10.1158/1078-0432.CCR-18-2984. Epub 2018 Nov 30. PMID 30504426
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Cabel L, Bonneau C, Bernard-Tessier A, Hequet D, Tran-Perennou C, Bataillon G, Rouzier R, Feron JG, Fourchotte V, Le Brun JF, Benoit C, Rodrigues M, Scher N, Minsat M, Legrier ME, Bieche I, Proudhon C, Sastre-Garau X, Bidard FC, Jeannot E. HPV ctDNA detection of high-risk HPV types during chemoradiotherapy for locally advanced cervical cancer. ESMO Open. 2021 Jun;6(3):100154. doi: 10.1016/j.esmoop.2021.100154. Epub 2021 May 19. PMID 34022731
- [Background] Jeannot E, Becette V, Campitelli M, Calmejane MA, Lappartient E, Ruff E, Saada S, Holmes A, Bellet D, Sastre-Garau X. Circulating human papillomavirus DNA detected using droplet digital PCR in the serum of patients diagnosed with early stage human papillomavirus-associated invasive carcinoma. J Pathol Clin Res. 2016 Jun 28;2(4):201-209. doi: 10.1002/cjp2.47. eCollection 2016 Oct. PMID 27917295
- [Background] Jeannot E, Latouche A, Bonneau C, Calmejane MA, Beaufort C, Ruigrok-Ritstier K, Bataillon G, Larbi Cherif L, Dupain C, Lecerf C, Popovic M, de la Rochefordiere A, Lecuru F, Fourchotte V, Jordanova ES, von der Leyen H, Tran-Perennou C, Legrier ME, Dureau S, Raizonville L, Bello Roufai D, Le Tourneau C, Bieche I, Rouzier R, Berns EMJJ, Kamal M, Scholl S. Circulating HPV DNA as a Marker for Early Detection of Relapse in Patients with Cervical Cancer. Clin Cancer Res. 2021 Nov 1;27(21):5869-5877. doi: 10.1158/1078-0432.CCR-21-0625. Epub 2021 Jul 1. PMID 34210686
- [Background] Lefevre AC, Pallisgaard N, Kronborg C, Wind KL, Krag SRP, Spindler KG. The Clinical Value of Measuring Circulating HPV DNA during Chemo-Radiotherapy in Squamous Cell Carcinoma of the Anus. Cancers (Basel). 2021 May 18;13(10):2451. doi: 10.3390/cancers13102451. PMID 34070045